CLINICAL TRIAL: NCT03298152
Title: One Year Clinical Evaluation of E-max CAD Versus Cerasmart Endocrowns in Anterior Endodontically Treated Teeth:A Randomized Clinical Trial
Brief Title: One Year Clinical Evaluation of E-max CAD Versus Cerasmart Endocrowns in Anterior Endodontically Treated Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Norhan Naief Abd El Haliem, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-09-29
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Endodontically Treated Teeth
Keywords: lithium disilicate endocrowns; cerasmart endocrowns
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emax CAD Endocrowns (Active Comparator): Using lithium disilicate e.max restorations is documented in literature as a successful restoration. Two different ceramic crowns systems were investigated clinically for three-years and howed that patient was satisfied with the final restoration
  Interventions: Procedure: Emax Endocrown
- Cerasmart Endocrowns (Experimental): A new material CERASMART (Force Absorbing Flexible nano ceramic CAD/CAM block) with high density of ultrafine glass particles with 71 wt% filled nano-composite. It combines high strength and unique aesthetics. full homogeneous and even distribution nano ceramic network lead to unique physical properties for cerasmart . Uniform scuttle (very short inter-particle distance) of silanated and bonded particles is key to delivering CERASMART's™ with exceptional strength, retention, acceptable level of marginal adaptation
  Interventions: Procedure: CERASMART Endocrown

INTERVENTIONS:
Procedure: CERASMART Endocrown — Endocrown fixed restoration used to restore endodontically treated anterior teeth using CERASMART blocks
  Arms: Cerasmart Endocrowns
Procedure: Emax Endocrown — Endocrown fixed restoration used to restore endodontically treated anterior teeth using Emax material
  Arms: Emax CAD Endocrowns

SUMMARY:
Nowadays Endocrowns are classified as conservative treatment modality for restoration of Endodontically treated teeth in which pulp chamber is used as a retentive resource.

With the advancement in technology in the field of adhesive dentistry its use is increasing day by day in clinical practice. Acid Etchable ceramics such as lithium Disilicate based ceramics are the gold standard ceramic material used for Endocrowns. The Etchable property and the translucent character of lithium Disilicate enhance strength and esthetic property.

A new material CERASMART (Force Absorbing Flexible nano ceramic CAD/CAM block) contain high density of ultrafine glass particles with 71 wt% filled nano-composite. It combines high strength and unique aesthetics. full homogeneous and even distribution of nano ceramic network lead to unique physical properties for cerasmart . Uniform scuttle (very short inter-particle distance) of silanated and bonded particles is key to delivering CERASMART's™ with high strength and acceptable level of marginal adaptation.

So, it can perfectly use in posterior, anterior, inlay, onlay, and implant restorations and also enables minimum tooth reduction for more conservative restoration.

Awad et al (1) found that Cerasmart showed significantly higher flexural strength and modulus of elasticity, with lower flexural modulus values compared to other groups. Also, result in smoother margins compared with other types of ceramic.

So, present research will evaluate patient satisfaction, bonding properties and marginal adaptation

DETAILED DESCRIPTION:
This study will carried out on patients collected from the dental clinics in fixed prosthodontics clinic, Faculty of Dentistry, Cairo University

the visits will be designed as follows:

.1st visit: (N.N) will call participants before tooth preparation procedure for X-ray reviewing and pre-operative photographing using a Professional digital camera also; Impression will be taken using the alginate impression material * for study cast analysis with suitable stock tray** size.

Each participant will be asked to sign consent form written in patient native language.

2nd visit: (Tooth preparation) After performing adequate disinfection and sterilization process for each instrument and tools will be used in this trial; the anesthetic solution (Anesthetic solution: Septanest SP, 4%, Septodont, France.) will be injected using infiltration technique. Then patients will be left from five to ten minutes then; the operator will check with the subjective for anasthesia.

Full preparation will be carried out following the principles of Endocrown preparation with deep chamfer finish line while 2 observers will select visually the appropriate shade. Final vinylpolysiloxane impressions will be taken for each participant in each groupusing the suitable tray size.

After final setting impressions will be checked for accuracy using magnifying loops (Magnifying loop: Univet optical technologies, Italy).

Then protemp temporary endocrowns ) Temporary crown material: Structure, Voco, GMBH, Germany.( will be cemented using eugenol free (Temporary cement: RelyX Temp, USA).

Impressions will be sent to the lab, poured with extra hard stone material. Then it will be removed from the impression after complete setting.

Endorowns for each patient will be fabricated using either lithium di-silicate material (Emax) or Cerasmart blocks according to the random allocation of the patients

3rd visit: Participants will be called again for final cementation. Temporary crown will be removed and abutments will be cleaned of any residues using pumice slurry ) Pumice slurry: DCL, Dental composite LTD, England.( applied with bristle brush and rubber cup under water irrigation.

Proper isolation will be done before cementation then permanent dual cure resin cement (Permanent cement: Bifix-QM, Voco Gmbh, Germany ) will be used for luting of permanent crowns according to manufacturer instructions. Ask the patients to hold the crown under occlusal compression until luting cement polymerization. 5 minutes later, excess cement will be removed.

Measuring of different outcomes will start in this visit for all patients.

The following assessment surveys (clinical evaluations) will done for both groups:

All patients will be recalled after 3, 6, 9, and 12 months. For each recall examination, evaluator will performed the direct clinical evaluation using modified USPHS criteria for margin integrity and gross fracture.

Visual inspection will be used for gross fracture evaluation. Endorowns that intact and fully retained will be rated 'Alfa', Endocrowns with partially retained with some portion of the restoration still intact will be rated as 'Bravo'and endocrowns completely missing will be rated as 'Charlie'.

Visual inspection and explorer will be using for marginal integrity evaluation. Endocrowns with no catch with The explorer and no visible crevice along the periphery of the restoration will be rated as Alpha (A), Endocrowns with explorer catches with visible evidence of a crevice, with and/or the base is not exposed, and the restoration is not mobile will be rated as Bravo (B) and endocrowms with explorer penetrates and extended to the dento-enamel junction will be rated as Charlie ©.

In addition, questionnaires will be used to evaluate patients' satisfaction and potential postoperative discomfort as the following questions:

1. Are you satisfied with your endocrown appearance?
2. Are you satisfied with your endocrown shade?
3. Do you feel your endocrown are poorly aligned?
4. Do you feel your endocrown are protruding?
5. Are you hiding your teeth while smiling?

Adherence improvement session will be taking place in the initial visit. This session will include:

* Each patient will be informed about the study steps and maintain oral hygiene. Subsequent sessions will occur at the follow-up visits.
* The patients will be trained for tooth brushing, flossing and instructed all oral hygiene methods after each meal.
* Instruct the patients to record any abnormalities or mobility in endocrowns.
* Recall appointment will be performed every two months for aduration of one year to stress on oral hygiene.
* Data collection methods:

Prosthodontic colleague will assess the outcome of each group. Data will be collected on excel sheets. All categorical data will be presented as risk ratios, while numerical data will be presented by mean and standard deviation. All data will be reported at a confidence interval of 95% and a p value of 5%.

Each factor will be measured as explained in the outcome table. - Outcome results will be written down on the patients' folders by (NN), then will be given to (JG) for data management. All the information will be transferred on excel sheets and saved on a computer in safe place and locked with a password only known to JG. A copy of the data will be saved on a flash drive with JG to provide a back up for the data.

Plans to increase participant retention & complete follow-up:

Telephone numbers of each patients and address will be taken and included in study, then phone calls and messages will be sent to remind patients before each appointment.

Data management:

JG will enter all data electronically. Patient files are to stored in numerical order in a secured place. J.G and A.Z will have access to data

Data Monitoring:

AZ will be responsible of data monitoring if any lost or delete occurs, in that case: back up data will be taken from (J.G) to provide hard copy for the requested data and A.Z will make final decision.

Harms:

If 50% of the patients showed any unfavorable signs as sever pain, irreparable fracture or shade changes which might affect the results. Then the treatment will be considered as stopped guidelines which necessitate stopping the treatment and interim analysis will be performed.

Auditing:

Auditing of the study design will be done by (AZ).

Ethics and dissemination Research ethics approval Protocol and informed consent form will be reviewed by the Ethics Committee of Scientific Research - faculty of Dentistry - Cairo University.

Protocol amendments:

Any changes in protocol affect the conduct of the study, benefit for patient or patient safety, including changes in study objectives, study design, sample size, study procedures, or significant administrative aspect will require formal amendment to the protocol. Such amendment will be agreed upon by the Council of Department of fixed prosthodontics, Faculty of Dentistry, Cairo University.

Consent:

Researcher will discuss the trial with all patients. Then patient can have an informed discussion with the researcher. Researcher will obtain written consent from patients willing to participate in the trial. All consent forms will write in Arabic language (Appendix 1.1).

Confidentiality:

All information related to study will store securely. All participants' information will store in locked cabinets in areas with limited access. To maintain participant confidentiality all data collection, process, and administrative forms will identify only by a coded ID number. All information related to patient names or other personal identifiers will store separately identified by code number. All local databases will be secured with password-protected access systems.

Access to data:

The investigator and supervisors will give access to the data sets. All data sets will be protected by password. To ensure confidentiality, Participant study information will become confidentially.

Ancillary and post-trial care:

All patients will be followed up 2 years even after the trial ends then might be used for further cohort study.

Dissemination policy:

o Study results will be published as partial fulfillment the Requirements for PHD degree in fixed prosthodontics.

ELIGIBILITY:
Inclusion Criteria:

- 1. Age range of the patients from 20-60 years old who can read and sign informed consent document.

2. Medically free patients or with controlled systemic disease. 3. No active periodontal disease.

Exclusion Criteria:

- 1. Patients under 20 years old. 2. Patients with bad oral hygiene and motivation. 3. Patients with psychiatric problems or unrealistic expectation (patient have phobia from dental treatments or needle bricks).

4. Patients with parafunctional habits (clencing/bruxism).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Gross Fracture | one year
  Categorical Alpha (A): Restoration is intact and fully retained.
  Bravo (B): Restoration is partially retained with some parts of the restoration still intact.
  Charlie (C): Restoration is completely missing

SECONDARY OUTCOMES:
Patient satisfaction | one year
  score by Visual Analogue Scale (VAS)
Marginal Integrity | one year
  Categorical Alpha (A): The explorer does not catch and no visible crevice along the periphery of the restoration.
  Bravo (B): The explorer catches and with visible evidence of a crevice, which the explorer penetrates, indicating that the edge of the restoration does not adapt closely to the tooth structure. Both dentin and/or the base is not exposed, and no mobility in the restoration.
  Charlie ©: The explorer penetrates and extended to the dento-enamel junction.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No